CLINICAL TRIAL: NCT00641680
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel-group, Phase IIIb Study to Assess the Efficacy, Safety & Product Attributes of Rhinocort Aqua(Budesonide) Versus Placebo and FluticasonePropionate as an Active Comparator in Patients 12yrs Age &Older With SeasonalAllergicRhinitis
Brief Title: Rhinocort Aqua Versus Placebo and Fluticasone Propionate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5360C00005
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Seasonal allergic rhinitis; Nasal symptoms; Congestion; Rhinorrhea; Sneeze; budesonide; Rhinocort AQUA; Fluticasone propionate; Flonase
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinorrhea; Sneezing | interventions — Budesonide; Fluticasone

ARMS (3):
- 1 (Experimental): Budesonide
  Interventions: Drug: Budesonide
- 2 (Active Comparator): Fluticasone propionate
  Interventions: Drug: Fluticasone propionate
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide
  Other Names: Rhinocort AQUA
  Arms: 1
Drug: Fluticasone propionate
  Other Names: Flonase®
  Arms: 2
Drug: Placebo
  Arms: 3

SUMMARY:
The purpose of this study is to compare once daily treatment with Rhinocort against placebo and Fluticasone Propionate at reliving the nasal symptoms of seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* At least a 2 year documented history of seasonal allergic rhinitis
* who, in the opinion of the investigator,
* is a candidate for treatment with nasal steroids based on a history of either

  * a)inadequate control of symptoms with antihistamines, decongestants and/or immunotherapy, or
  * b) prior successful treatment with nasal steroids.
* A positive response to a skin prick test at Visit 1 or within the last 12 months for grass allergens that must be present in the subject's environment for the duration of the study.

Exclusion Criteria:

* Primary or secondary adrenal insufficiency
* Nasal candidiasis, rhinitis medicamentosa, acute or chronic sinusitis, influenza, upper respiratory tract infection or structural abnormalities of the nose (e.g., septal deviation, nasal polyps) symptomatic enough to cause significant nasal obstruction as judged by the investigator.
* A diagnosis of asthma requiring treatment as specifies in the protocol.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2003-04; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
To compare once daily treatment with Rhinocort against placebo and at reliving the nasal symptoms of seasonal allergic rhinitis. | 2 weeks

SECONDARY OUTCOMES:
To compare once daily treatment with Rhinocort against Fluticasone Propionate at reliving the nasal symptoms of seasonal allergic rhinitis. | 2 weeks
To compare once daily treatment with placebo against Fluticasone Propionate at reliving the nasal symptoms of seasonal allergic rhinitis. | 2 weeks
Safety assessment via adverse events and clinical measurements. | 2 & 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Ruff, MD, Principal Investigator — Pharmaceutical Research, Dallas, USA